CLINICAL TRIAL: NCT06466772
Title: Precision Sensorimotor Neurorehabilitation Through Personalized Stimulation Loops
Acronym: StimuLOOP-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Switzerland) (Other); Cereneo AG (Industry); University Children's Hospital, Zurich (Other); Vontobel-Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-01194
Record Dates: First submitted 2024-04-11; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Consolidation arm: hyper-personalized feedback-based motor rehabilitation with targeted auditory stimulation during sleep (HPF intervention, TASS intervention)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptation arm (Sham Comparator): Hyper-personalized feedback-based motor rehabilitation with sham targeted auditory stimulation during sleep (HPF intervention, TASS sham intervention)
  Interventions: Behavioral: Hyper-personalized feedback (HPF intervention); Behavioral: Control targeted auditory stimulation during sleep (TASS sham intervention)
- Consolidation arm (Experimental): Hyper-personalized feedback-based motor rehabilitation with targeted auditory stimulation during sleep (HPF intervention, TASS verum intervention)
  Interventions: Behavioral: Hyper-personalized feedback (HPF intervention); Behavioral: Targeted auditory stimulation during sleep (TASS verum intervention)

INTERVENTIONS:
Behavioral: Hyper-personalized feedback (HPF intervention) — For lower limb motor rehabilitation, the investigator will employ real-time continuous feedback for movement aspects that are specific to each participant's motor deficit. The feedback will be adapted and tailored to each participant.
Behavioral: Targeted auditory stimulation during sleep (TASS verum intervention) — The investigator aim to reactivate rehabilitation- related memories through the presentation of auditory stimuli during sleep with the goal of promoting motor memory consolidation into stable motor commands
  Arms: Consolidation arm
Behavioral: Control targeted auditory stimulation during sleep (TASS sham intervention) — Identical auditory presentation during the motor rehabilitation training, but not during the night (sham promotion memory reactivation)
  Arms: Adaptation arm

SUMMARY:
Stroke is the most common neurological disease in the elderly population and accounts for substantial disability and health care costs. Disability is largely driven by mobility deficits caused by impaired gait. Effective treatments are available to restore lower limb function and improve gait, but response to treatment varies greatly from patient to patient and often shows only small effect sizes. Addressing this heterogeneity requires personalization, a concept referred to precision neurorehabilitation.

StimuLOOP.S intends to foster structured and reproducible methods for precision neurorehabilitation of gait in stroke. The investigator will carry out a proof-of-concept study to investigate the integration of two personalized methods for each patient. Two innovative technologies are applied in concert to enhance the recovery of lower limb function.

1. Hyper-personalized feedback (HPF): For lower limb motor rehabilitation, the investigator will employ real-time continuous feedback for movement aspects that are specific to each participant's motor deficit. The feedback will be adapted and tailored to each participant. This results in a two-step personalization; in the first step, the investigator will choose what movement aspect is therapeutically targeted, and in the second step, the investigator will define the feedback presented to the participant.
2. Targeted auditory stimulation during sleep (TASS):The investigator aim to reactivate rehabilitation- related memories through the presentation of auditory stimuli during sleep with the goal of promoting motor memory consolidation into stable motor commands.

The HPF intervention is expected to induce rapid adaptations, which however do not persist over multiple days. To counter this, the investigator will leverage memory reactivation during sleep to enhance the consolidation of the movement patterns that are learned during HPF.

The investigator expect that these interventions will lead to greater gains in functional walking ability. Beyond demonstrating a proof-of-concept for novel methods of precision neurorehabilitation, positive results of this project may have implications for neurorehabilitation treatment in general by providing first insights into the benefits and interplay of HPF and TASS.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or intracerebral hemorrhage with a gait deficit older than 30 days but not more than 6 months.
* Functional Ambulation Category ≥3
* ≥18 years of age
* Informed consent as documented by signature

Exclusion Criteria:

* Cognitive impairment, Montreal Cognitive Assessment (MoCa) < 20
* Comprehensive aphasia precluding the understanding of study-related information
* Previous stroke that caused sustained clinically relevant cognitive, visual and/or gait deficits
* Expected acute hospitalization during the training period
* History of a physical or neurological condition that interferes with study procedures
* Social and/or personal circumstances that interfere with the ability to return for therapy sessions and follow-up assessments
* Not capable of voluntary gait adaptation
* Allergy to nickel
* Patients taking benzodiazepines or Z-drugs with a significant effect on sleep EEG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
6 min walking test (6MWT) | Pre, immediately post motor rehabilitation training and one-month post-training
  Change in functional walking ability assessed with the 6 min walking test (6MWT)

SECONDARY OUTCOMES:
Gait kinematics | Pre, immediately post motor rehabilitation training and during 15 days of motor rehabilitation training and one-month post-training
  Motor learning assessed via changes in gait kinematics: variability, symmetry, coordination, stability.

OTHER OUTCOMES:
Single-channel sleep EEG (Electroencephalography)+ EMG (Electroencephalography) + EOG (Electrooculography) | During 15 days of motor rehabilitation training
  Single-channel sleep EEG (Electroencephalography): sleep architecture, ERSP, ERP, frequency spectrum, slow-wave activity changes, changes in the spindle band, sleep oscillation detection (K-complexes, spindles, slow-wave-spindle-coupling)
  EMG ( Electromyography): signal from the chin recorded during sleep will be filtered between 10 and 100 Hz and re-referenced bilaterally according to AASM criteria and used for offline sleep staging
  EOG (Electrooculography): filtered between 0.3 and 35 Hz and used for offline sleep staging.
  EOG and EMG are only used for sleep scoring
Sleep hdEEG + EMG + EOG | Pre motor rehabilitation training
  Sleep high density EEG: sleep architecture, slow-wave activity topography, spindle band topography, ERSP, ERP, frequency spectrum, sleep oscillation detection (K-complexes, spindles, slow-wave-spindle-coupling).
  EOG (Electrooculography)and EMG ( Electromyography) are only used for sleep scoring
Wake hdEEG | Pre and immediately post motor rehabilitation training
  Wake high density EEG: theta topography, alpha topography, frequency spectrum at resting state, ERP in oddball task, ERSP in oddball task, characterization of wake slow waves if detectable
Quality of Life (EQ-5D-5L) | Pre motor rehabilitation training and 1 month after training
  Patient-Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No